CLINICAL TRIAL: NCT01758718
Title: Eyelash Line Resection for Entropion Associated With Down's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Associate professor of Ophthalmology, Kyorin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kyorineye009; Entropion with Down's syndrome
Record Dates: First submitted 2012-12-27; First posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-12

CONDITIONS: Down's Syndrome
Keywords: Down's syndrome; entropion; lid plasty
MeSH Terms: conditions — Down Syndrome; Entropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Entropion with Down's syndrome (Active Comparator): Eyelash resection surgery was performed for entropion with Down's syndrome
  Interventions: Procedure: Eyelash line resection

INTERVENTIONS:
Procedure: Eyelash line resection — Eyelash resection surgery was performed for entropion with Down's syndrome
  Other Names: Lid plastic surgery

SUMMARY:
Surgical outcome of entropion associated with Down's syndrome was evaluated. Grading scale of superficial punctate keratopathy and score of wearing glasses to correct refractive errors were measured.

ELIGIBILITY:
Inclusion Criteria:

* The patients with entropion with Down's syndrome

Exclusion Criteria:

* The patients of Down's syndrome who do not have entropion.

Ages: 3 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Grading scale of superficial punctate keratopathy | one year
  The degree of superficial punctate keratopathy was assessed by the area and density classification which was scored with the area of superficial punctate keratopathy graded from A0 through A3, and the density graded from D0 through D3.

SECONDARY OUTCOMES:
Score of wearing glasses | one ear
  The score of wearing glasses was graded 2; all day, 1; more than half day, 0; none of the day.

CONTACTS AND LOCATIONS:
Overall Officials: Akito Hirakata, MD, Study Chair — Kyorin Eye Center
Locations (1):
- Kyorin Eye Center, Mitaka, Tokyo, Japan

REFERENCES:
- [Derived] Suzuki Y, Hama Y, Yoshikawa-Kobayashi I, Tomita K, Inoue M, Hirakata A. Eyelash line resection for cilial entropion in patients with Down's syndrome. Br J Ophthalmol. 2014 Oct;98(10):1442-7. doi: 10.1136/bjophthalmol-2014-304946. Epub 2014 May 15. PMID 24831720